CLINICAL TRIAL: NCT06377488
Title: Evaluation of the Clinical Performance of Daily Disposable Silicone Hydrogel Multifocal Toric Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-6542
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Results first posted 2025-07-09 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Visual Acuity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Test Arm (Experimental): Eligible subjects who are habitual soft contact lens wearers will be fit with the TEST lens in both eyes, to wear the lens for a minimum of 6 hours a day, every day, between visits for approximately 2 weeks.
  Interventions: Device: JJVC Investigational Multifocal Toric Contact Lens manufactured in Senofilcon A (C3) material with UV blocker / HEV filter

INTERVENTIONS:
Device: JJVC Investigational Multifocal Toric Contact Lens manufactured in Senofilcon A (C3) material with UV blocker / HEV filter — Test Lens

SUMMARY:
This will be an open-label, 3-visit, single-arm, dispensing clinical trial to evaluate visual acuity.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be at least 40 and not more than 70 years of age at the time of screening.
4. Own a wearable pair of spectacles if required for their distance vision.
5. Be an adapted soft contact lens wearer in both eyes (i.e. worn lenses for at least 8 hours per day at least two days per week for the past 4 weeks).
6. Be already wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".
7. The subject's distance spherical component of their refraction must be in the range of either -1.25 D to -3.75 D, or +1.25 D to +4.25 D.
8. The subject's refractive cylinder must be in the range of -1.00 D to -1.75 D in each eye, with the cylinder axes in the range of either 90°±15° or 180°±15°.
9. The subject's ADD power must be in the range of +0.75 D to +2.50 D in each eye.
10. The subject must have best corrected distance visual acuity of 20/20-3 or better in each eye.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

The subject must not:

1. Be currently pregnant or lactating.
2. By self-report, have any systemic disease (e.g. Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis), or other diseases, which are known to interfere with contact lens wear and/or participation in the study.
3. Use systemic medications that may interfere with contact lens wear or cause blurred vision. See Section 9.1 for additional details regarding excluded systemic medications.
4. Currently use ocular medication (with the exception of rewetting drops).
5. Have any known hypersensitivity or allergic reaction to single use preservative free rewetting drops or sodium fluorescein.
6. Have had any previous, or have any planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, cataract surgery, retinal surgery, etc.).
7. Have had previous eyelid injuries, surgeries or procedures which are known to have caused abnormal eyelid position or movement, by self-report.
8. Have participated in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.
9. Be an employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
10. Have a history of amblyopia or strabismus, by self-report.
11. Have a history of herpetic keratitis, by self-report.
12. Have ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion.
13. Have any Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA scale.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (15):
- United States (15):
  - Dr. James Weber & Associates, PA - City Square Blvd, Jacksonville, Florida
  - Stam & Associates Eye Care, Jacksonville, Florida
  - Omega Vision Center, Longwood, Florida
  - Maitland Vision Center - North Orlando Ave, Maitland, Florida
  - Mid-State Eye, Clinton, Illinois
  - Kannarr Eye Care, Pittsburg, Kansas
  - Birmingham Vision Care, Bloomfield Hills, Michigan
  - Center for Ophthalmic and Vision Research/Eye Associates of New York, Manhattan, New York
  - Sacco Eye Group, Vestal, New York
  - ProCare Vision Centers, Granville, Ohio
  - Luxe Vision and Optical, Powell, Ohio
  - Dr. David W. Ferris & Associates, Warwick, Rhode Island
  - Optometry Group, LLC, Memphis, Tennessee
  - Tyler Eye Associates, Tyler, Texas
  - New River Vision Care, Oak Hill, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 176 subjects were enrolled in this study. Of those enrolled, 171 subjects were dispensed the study lens, while 5 subjects failed to meet all eligibility criteria. Of those dispensed, 163 subjects completed the study while 8 subjects were discontinued.
Groups:
- Test (Senofilcon A C3): Subject that wore the Test lens at any point during the study.
Period: Overall Study
Arm/Group | Test (Senofilcon A C3)
Started | 171
Completed | 163
Not Completed | 8
Not completed — Unsatisfactory Visual Response due to Test Article | 2
Not completed — Unsatisfactory Lens Fitting due to Test Article | 2
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 1
Not completed — Incorrect Lens Dispensed | 2

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens.
Groups:
- Myopes: Subjects were classified as Myopic if the distance spherical equivalent refraction was in the range of -1.25 D to -3.75 D.
- Hyperopes: Subjects were classified as Hyperopic if the distance spherical equivalent refraction was in the range of +1.25 D to +4.25 D.
- Total: Total of all reporting groups
Arm/Group | Myopes | Hyperopes | Total
Number analyzed (Participants) | 105 | 66 | 171
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (6.89) | 59.1 (6.10) | 53.5 (7.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 51 | 119
  Male | 37 | 15 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 9 | 3 | 12
  White | 93 | 62 | 155
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 105 | 66 | 171

OUTCOME MEASURES:

1. Primary Outcome: HLHC Binocular logMAR Visual Acuities
Description: Binocular visual acuity was measured on a logMAR (Logarithm of Minimal Angle of Resolution) scale under high luminance high contrast condition. At distance (4 meters), VA is assessed using ETDRS (Early Treatment Diabetic Retinopathy Study) charts; while near (40 cm) and intermediate (64 cm) assessments were made using reduced Guillon-Poling charts. Letter-by-letter results calculated the visual performance score for each chart read. LogMAR scores closer to zero, or below zero, indicate a better visual acuity. A logMAR visual performance score of 0.0 is equivalent to Snellen visual acuity of 20/20. Data from hyperopes and myopes were combined for this outcome since logMAR scores between the two populations are similar.
Time Frame: 2-Week Follow-up
Population: All dispensed subjects regardless of deviation from protocol with data collected at the 2-week follow-up.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Test (Senofilcon A C3)
Number analyzed (Participants) | 163
logMAR
  Distance (4m) | -0.088 (0.0874)
  Intermediate (64cm) | -0.018 (0.1106)
  Near (40cm) | 0.087 (0.1103)
Statistical Analysis 1: Comparison: Test (Senofilcon A C3); It was calculated using a 1-sided one-sample mean t-test with a family wise type I error rate of 5% with at least 99% statistical power, that 9, 6 and 29 subjects were required to test the primary hypotheses for distance, intermediate and near, respectively; Test type: Superiority; Mixed Model Analysis; The Satterthwaite Method was used for the calculation of the denominator degrees of freedom; least-square mean estimate = -0.085, 95% CI 2-sided [-0.115 to -0.056], Standard Error of Mean 0.0139 — Visual Acuity scores at distance was estimated using 95% confidence intervals (CI) constructed for the least-square mean (LSM)
Statistical Analysis 2: Comparison: Test (Senofilcon A C3); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mixed Model Analysis; The Satterthwaite Method was used for the calculation of the denominator degrees of freedom; least-square mean estimate = -0.023, 95% CI 2-sided [-0.050 to 0.005], Standard Error of Mean 0.0131 — Visual Acuity scores at intermediate was estimated using 95% confidence intervals (CI) constructed for the least-square mean (LSM)
Statistical Analysis 3: Comparison: Test (Senofilcon A C3); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mixed Model Analysis; The Satterthwaite Method was used for the calculation of the denominator degrees of freedom; least-square mean estimate = 0.083, 95% CI 2-sided [0.051 to 0.116], Standard Error of Mean 0.0152 — Visual Acuity scores at near was estimated using 95% confidence intervals (CI) constructed for the least-square mean (LSM)

2. Primary Outcome: CLUE Vision Scores
Description: Subjective vision was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE vision score for each sphere stratum (Hyperope and Myope) was reported.
Time Frame: 2-Week Follow-up
Population: All dispensed subjects regardless of deviation from protocol with data collected at the 2-week follow-up.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Test (Senofilcon A C3)
Number analyzed (Participants) | 164
Units on a Scale
  Myopes: number analyzed (Participants) | 101
  Myopes | 61.13 (21.181)
  Hyperopes: number analyzed (Participants) | 63
  Hyperopes | 56.19 (18.634)
Statistical Analysis 1: Comparison: Test (Senofilcon A C3); It was calculated using a 1-sided one-sample mean t-test with a family wise type I error rate of 5% with at least 99% statistical power, that 23 and 29 subjects were required to test for superiority for CLUE vision scores for hyperopes and myopes, respectively; Test type: Superiority; Mixed Model Analysis; The Satterthwaite Method was used for the calculation of the denominator degrees of freedom; Mean Population Estimate = 62.1, 95% CI 2-sided [56.7 to 67.5], Standard Error of Mean 2.6 — Mean estimates were conducted for myopes only using two-sided confidence intervals (CI) constructed for the least square mean
Statistical Analysis 2: Comparison: Test (Senofilcon A C3); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Mixed Model Analysis; The Satterthwaite Method was used for the calculation of the denominator degrees of freedom; Mean Population Estimate = 57.8, 95% CI 2-sided [51.7 to 64.0], Standard Error of Mean 3.02 — Mean estimates were conducted for hyperopes only using two-sided confidence intervals (CI) constructed for the least square mean

3. Primary Outcome: Proportion of Eyes With Absolute Rotation Less Than or Equal to 10 Degrees
Description: Absolute rotation was assessed for each subject eye using a slit lamp 15-minutes after lens insertion. Acceptable absolute rotation was dichotomized into a binary response where Y=1 if absolute rotation was less than or equal to 10 degrees and Y=0 otherwise (absolute rotation greater than 10 degrees). The proportion of eyes with absolute rotation less than or equal to 10 degrees was report for each lens.
Time Frame: 15-minutes after lens insertion
Population: All dispensed subjects regardless of subsequent withdrawal from study or deviation from protocol.
Measure: Number; unit: Proportion of eyes
Units Other Than Participants: Eyes
Arm/Group | Test (Senofilcon A C3)
Number analyzed (Participants) | 171
Number analyzed (Eyes) | 342
Proportion of eyes | 0.9474
Statistical Analysis 1: Comparison: Test (Senofilcon A C3); It was calculated using a Bayesian beta-binomial model for correlated data with a reference rate of 0.902 and an intraclass correlation of 0.70, that 140 subjects were required to test for superiority to achieve a minimum statistical power of 96% with 95% central posterior credible interval; Test type: Superiority; Bayesian beta-binomial model; Bayesian beta-binomial model with correlated binary data; Central Posterior Mean Estimate = 0.943, 95% CI 2-sided [0.908 to 0.968], Standard Deviation 0.0155

4. Primary Outcome: Proportion of Eyes With Rotational Stability Less Than or Equal to 5 Degrees
Description: Rotational Stability was assessed for each subject eye using a slit lamp 15-minutes after lens insertion. Rotational Stability was dichotomized into a binary response where Y=1 if Rotational Stability was less than or equal to 5 degrees and Y=0 otherwise (Rotational Stability greater than 5 degrees). The proportion of eyes with Rotational Stability less than or equal to 5 degrees was report for each lens.
Time Frame: 15-minutes after lens insertion
Population: All dispensed subjects regardless of subsequent withdrawal from study or deviation from protocol.
Measure: Number; unit: Proportion of eyes
Units Other Than Participants: Eyes
Arm/Group | Test (Senofilcon A C3)
Number analyzed (Participants) | 171
Number analyzed (Eyes) | 342
Proportion of eyes | 1
Statistical Analysis 1: Comparison: Test (Senofilcon A C3); It was calculated using a Bayesian beta-binomial model for correlated data with a reference rate of 0.99 and an intraclass correlation of 0.70, that 140 subjects were required to test for superiority to achieve a minimum statistical power of 96% with 95% central posterior credible interval; Test type: Superiority; Bayesian beta-binomial model; Bayesian beta-binomial model with correlated binary data; Central Posterior Mean Estimate = 0.988, 95% CI 2-sided [0.974 to 0.997], Standard Deviation 0.0058

5. Primary Outcome: Proportion of Eyes With Grade 3 or Higher Slit Lamp Findings
Description: Slit Lamp Findings (SLF) were assessed using a biomicroscope and was graded using the FDA grading scale (Grade: 0, 1,2, 3 and 4) with grade 0 represents the absence of findings and 1 to 4 representing successively worse findings (i.e. Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe). This was performed on each subject eye at every study visit (baseline, unscheduled visits and 1-week follow-up). The data was then dichotomized into two groups. Those with grade 3 or higher and those with grade 2 or lower. The proportion of eyes with SLF with grade 3 or higher was reported. Data from the hyperope and myopes group were combined for this outcome since the rate of SFLs grade 3+ is similar for these two populations.
Time Frame: Up to 2-Week Follow-up
Population: All dispensed subjects regardless of subsequent withdrawal from study or deviation from protocol.
Measure: Number; unit: Proportion of eyes
Units Other Than Participants: Eyes
Arm/Group | Test (Senofilcon A C3)
Number analyzed (Participants) | 171
Number analyzed (Eyes) | 342
Proportion of eyes | 0.0029
Statistical Analysis 1: Comparison: Test (Senofilcon A C3); It was calculated that 140 subjects were required to test for superiority to achieve a minimum statistical power of 99% with 95% central posterior credible; Test type: Superiority; Bayesian beta-binomial model; Bayesian beta-binomial model with correlated binary data; Central Posterior Mean Estimate = 0.006, 95% CI 2-sided [0.000 to 0.017], Standard Deviation 0.0047

6. Primary Outcome: Proportion of Eyes With Unacceptable Lens Fitting
Description: Contact lens fitting acceptance was assessed for each subject eye using a biomicroscope post lens insertion at the 1-week follow-up.
  Lens fit was a binary variable where unacceptable lens fit=1 and acceptable lens fit=0. The proportion of eyes with unacceptable lens fit was reported. Data from the hyperope and myopes group were combined for this outcome since lens fitting characteristics are similar for these two populations.
Time Frame: Up to 2-Week Follow-up
Population: All dispensed subjects regardless of subsequent withdrawal from study or deviation from protocol.
Measure: Number; unit: Proportion of eyes
Units Other Than Participants: Eyes
Arm/Group | Test (Senofilcon A C3)
Number analyzed (Participants) | 171
Number analyzed (Eyes) | 342
Proportion of eyes | 0
Statistical Analysis 1: Comparison: Test (Senofilcon A C3); [analysis description as in outcome 5, analysis 1]; Test type: Superiority; Bayesian beta-binomial model; Bayesian beta-binomial model with correlated binary data; Central Posterior Mean Estimate = 0.003, 95% CI 2-sided [0.000 to 0.011], Standard Deviation 0.0029

7. Secondary Outcome: CLUE Vision Scores
Description: as for outcome 2
Time Frame: 2-Week Follow-up
Population: All dispensed subjects regardless of deviation from protocol with data collected at the 2-week follow-up.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Test (Senofilcon A C3)
Number analyzed (Participants) | 164
Units on a Scale
  Myopes: number analyzed (Participants) | 101
  Myopes | 61.13 (21.181)
  Hyperopes: number analyzed (Participants) | 63
  Hyperopes | 56.19 (18.634)
Statistical Analysis 1: Comparison: Test (Senofilcon A C3); It was calculated using a one-sided one-sample mean t-test with a family wise type I error rate of 5% with at least 99% statistical power, that 42 and 55 subjects were required to test for superiority for CLUE vision scores for hyperopes and myopes, respectively; Test type: Superiority; Mixed Model Analysis; The Satterthwaite Method was used for the calculation of the denominator degrees of freedom; Least-square mean estimate = 57.8, 95% CI 2-sided [51.7 to 64.0], Standard Error of Mean 3.02 — This is the analysis for hyperopes only. Mean estimates were conducted using two-sided confidence intervals (CI) constructed for the least square mean
Statistical Analysis 2: Comparison: Test (Senofilcon A C3); [analysis description as in outcome 7, analysis 1]; Test type: Superiority; Mixed Model Analysis; The Satterthwaite Method was used for the calculation of the denominator degrees of freedom; Least-square mean estimate = 62.1, 95% CI 2-sided [56.7 to 67.5], Standard Error of Mean 2.6 — This is the analysis for myopes only. Mean estimates were conducted using two-sided confidence intervals (CI) constructed for the least square mean

8. Secondary Outcome: CLUE Comfort Scores
Description: Subjective comfort was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE comfort scores for each sphere stratum (Hyperope and Myope) were reported.
Time Frame: 2-Week Follow-up
Population: All dispensed subjects regardless of deviation from protocol with data collected at the 2-week follow-up.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Test (Senofilcon A C3)
Number analyzed (Participants) | 164
Units on a Scale
  Myopes: number analyzed (Participants) | 101
  Myopes | 63.63 (22.498)
  Hyperopes: number analyzed (Participants) | 63
  Hyperopes | 62.56 (20.732)
Statistical Analysis 1: Comparison: Test (Senofilcon A C3); It was calculated using a one-sided one-sample mean t-test with a family wise type I error rate of 5% with at least 99% statistical power, that 23 and 46 subjects were required to test for superiority for CLUE comfort scores for hyperopes and myopes, respectively; Test type: Superiority; Mixed Model Analysis; The Satterthwaite Method was used for the calculation of the denominator degrees of freedom; Mean Population Estimate = 64.7, 95% CI 2-sided [58.6 to 70.8], Standard Error of Mean 3.02 — Mean estimates were conducted for hyperopes using two-sided confidence intervals (CI) constructed for the least square mean
Statistical Analysis 2: Comparison: Test (Senofilcon A C3); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; Mixed Model Analysis; The Satterthwaite Method was used for the calculation of the denominator degrees of freedom; Mean Population Estimate = 64.2, 95% CI 2-sided [59.0 to 69.5], Standard Error of Mean 2.54 — Mean estimates were conducted for myopes using two-sided confidence intervals (CI) constructed for the least square mean

9. Secondary Outcome: CLUE Handling Scores
Description: Subjective handling was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE handling scores for each sphere stratum (Hyperope and Myope) were reported.
Time Frame: 2-Week Follow-up
Population: All dispensed subjects regardless of deviation from protocol with data collected at the 2-week follow-up.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Test (Senofilcon A C3)
Number analyzed (Participants) | 164
Units on a Scale
  Myopes: number analyzed (Participants) | 101
  Myopes | 68.03 (19.455)
  Hyperopes: number analyzed (Participants) | 63
  Hyperopes | 67.88 (20.677)
Statistical Analysis 1: Comparison: Test (Senofilcon A C3); It was calculated using a one-sided one-sample mean t-test with a family wise type I error rate of 5% with at least 99% statistical power, that 15 and 26 subjects were required to test for superiority for CLUE handling scores for hyperopes and myopes, respectively; Test type: Superiority; Mixed Model Analysis; The Satterthwaite Method was used for the calculation of the denominator degrees of freedom; Mean Population Estimate = 67.9, 95% CI 2-sided [62.2 to 73.5], Standard Error of Mean 2.79 — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Test (Senofilcon A C3); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; Mixed Model Analysis; The Satterthwaite Method was used for the calculation of the denominator degrees of freedom; Mean Population Estimate = 67, 95% CI 2-sided [62.2 to 71.8], Standard Error of Mean 2.32 — [estimate comment as in outcome 8, analysis 2]

10. Secondary Outcome: Proportion of Subject Achieving Optimal Lens Pair in 4 Lenses or Less.
Description: The number of lenses to achieve the optimal pair for each subject was calculated as the original pair (2) plus all the required modifications to reach the optimal pair. In this study the minimum number of lenses per subject used was 2 where the maximum possible number of lenses used was 10. The data was dichotomized as Y=1 if the subject was able to achieve optimal lens pair in 4 lenses or lenses or less and 0 otherwise. A lens modification was performed if the subject reports unsatisfactory vision or was unable to obtain 20/30 distance visual acuity in both eyes. If the subject reported satisfactory vision with the lenses a modification was not required. However, based upon the investigator's findings on the measured visual acuity and/or over- refraction a modification may have been performed. Data for the hyperope and myope groups were combined for this endpoint since the number of subjects needed to optimize vision is independent of which group a subject belongs to.
Time Frame: Up to 1-Week Follow-up
Population: All dispensed subjects regardless of subsequent withdrawal from study or deviation from protocol.
Measure: Number; unit: Proportion of Subjects
Arm/Group | Test (Senofilcon A C3)
Number analyzed (Participants) | 171
Proportion of Subjects | 0.971
Statistical Analysis 1: Comparison: Test (Senofilcon A C3); It was calculated using a Bayesian beta-binomial model for correlated data with a reference rate of 0.99 and an intraclass correlation of 0.70 with 5000 replicating trials, that 140 subjects were required to test for superiority to achieve a minimum statistical power of 99% with 95% central posterior credible; Test type: Superiority; Bayesian beta-binomial model; Bayesian beta-binomial model with correlated binary data; Central Posterior Mean Estimate = 0.966, 95% CI 2-sided [0.933 to 0.988], Standard Deviation 0.0135

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; approximately 3 weeks per subject.
Description: All subjects dispensed the study lens.
Arm/Group | Test (Senofilcon A C3)
All-Cause Mortality (participants affected / at risk) | 0/171
Serious Adverse Events (participants affected / at risk) | 0/171
Other Adverse Events (participants affected / at risk) | 0/171

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT06377488/Prot_SAP_000.pdf